CLINICAL TRIAL: NCT00584805
Title: A Multi-Site Phase 2 Open-Label, Safety and Immunogenicity Study of Eastern Equine Encephalitis Vaccine, Inactivated, Dried, TSI-GSD 104 in Healthy Adults At Risk for Exposure to Eastern Equine Encephalitis Virus
Brief Title: Safety and Immunogenicity Study of Eastern Equine Encephalitis (EEE) Vaccine
Acronym: EEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-14568; FY06-31 (Other: SIP); S-09-12 (Other: Sponsor number)
Record Dates: First submitted 2007-12-19; First posted 2008-01-02 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2018-10

CONDITIONS: Eastern Equine Encephalitis
Keywords: EEE
MeSH Terms: conditions — Encephalomyelitis, Eastern Equine | interventions — Desiccation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccination (Experimental): Inactivated, Dried, TSI-GSD 104, EEE
  Interventions: Biological: Inactivated, Dried, TSI-GSD 104, EEE

INTERVENTIONS:
Biological: Inactivated, Dried, TSI-GSD 104, EEE — Subjects will receive 0.5ml SQ, as a two-dose primary series (days 0 and 28) and 0.1ml, as a mandatory booster dose at 6 months. A booster dose may be administered before 6 months if PRNT80 is < 1:40 after day 28. Up to four booster doses may be given in any 1-year period.
  Other Names: EEE A-14568

SUMMARY:
This study is designed to determine the safety and immunogenicity of Eastern Equine Encephalitis (EEE) Vaccine.

DETAILED DESCRIPTION:
This was an open-label, vaccine study of Eastern Equine Encephalitis Vaccine, Inactivated Dried, EEE, TSI-GSD 104 in healthy, adult subjects. No concurrent control group was used. The controls used in this study to assess immunogenicity were historical PRNT80 values obtained in past studies of the EEE vaccine. Rates of adverse events (AEs) were tabulated by relationship to product administration and severity.

The primary objectives are to assess the safety of Eastern Equine Encephalitis Vaccine, Inactivated, Dried EEE, TSI GSD 104, and to assess immunogenicity of Eastern Equine Encephalitis Vaccine, Inactivated, Dried EEE, TSI GSD 104.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* EEE PRNT80 ≤ 1:20.
* EEE PRNT80 ≤ 1:40 for booster series
* (females) Negative pregnancy test on the same day before vaccination.
* Not planning pregnancy for 3 months.
* At risk for exposure to virulent EEE virus (with up-to-date risk assessment).
* Up-to-date (within 1 year) physical examination/tests.
* Sign and date the approved informed consent.
* Willing to return for all follow-up visits.
* Agree to report adverse events (AE) up to 28 days after each vaccination.

Exclusion Criteria:

* Over 65 years of age (for Primary Immunization).
* Clinically significant abnormal lab results including evidence of Hepatitis C, Hepatitis B carrier state, or elevated (2X normal) liver function tests.
* History of immunodeficiency or current treatment with immunosuppressive medication.
* (females) Currently breastfeeding.
* Confirmed human immunodeficiency virus (HIV) titer.
* Any known allergies to components of the vaccine.
* A medical condition that, in the judgment of the Principal Investigator (PI), would impact subject safety (i.e.-vaccination or exposure to another Alphavirus).
* Administration of any IND product or live vaccine within 28 days of EEE.
* Any unresolved AEs resulting from a previous immunization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-06-03 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rivard, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- U.S. Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States

REFERENCES:
- [Derived] Schultz JS, Sparks H, Beckham JD. Arboviral central nervous system infections. Curr Opin Infect Dis. 2021 Jun 1;34(3):264-271. doi: 10.1097/QCO.0000000000000729. PMID 33899755

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 138 subjects were enrolled at Special Immunizations Clinic, Division of Medicine, U.S. Army Medical Research Institute of Infectious Diseases (USAMRIID), Fort Detrick, MD
Period: Overall Study
Arm/Group | Vaccination
Started | 138
Completed | 39
Not Completed | 99
Not completed — No longer at risk of exposure | 39
Not completed — Relocation | 36
Not completed — Withdrawal by Subject | 18
Not completed — Non-compliance | 1
Not completed — Lost to follow up | 3
Not completed — Screen failures | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vaccination
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: Years of age] | 39.0 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : White | 126
  Race : Black or African American | 3
  Race : Asian | 5
  Race : Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 138

OUTCOME MEASURES:

1. Primary Outcome: Subject Response Rates for PRNT80 Titers
Description: Subject response rates for PRNT80 titers for vaccinations and all boosters. The per-protocol population was used for immunogenicity analyses. Only subjects who were vaccinated according to the schedule defined in the protocol were included in the per-protocol population. Only observations or specimens collected according to the protocol were included in the analyses using the per protocol population. If a subject received one or more treatments out of compliance with the protocol schedule, any observations or specimens collected after the out-of-compliance treatment were excluded from the analyses using the per-protocol population.
  Four to 5 weeks for primary vaccinations (3) and up to four boost doses in 1 year period for a total duration of up to 5 years (anticipated duration of study execution).
Time Frame: 5 years
Population: Only observations or specimens collected according to the protocol were included in the analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination
Number analyzed (Participants) | 138
Participants
  Post dose 2: Day 21-35: number analyzed (Participants) | 65
  Post dose 2: Day 21-35 | 39
  Pre-month 6: number analyzed (Participants) | 61
  Pre-month 6 | 28
  Post month 6, Day 21-35: number analyzed (Participants) | 57
  Post month 6, Day 21-35 | 48
  Post booster 1, Day 21-35: number analyzed (Participants) | 102
  Post booster 1, Day 21-35 | 79
  Post booster 2, Day 21-35: number analyzed (Participants) | 38
  Post booster 2, Day 21-35 | 24
  Post booster 3, Day 21-35: number analyzed (Participants) | 19
  Post booster 3, Day 21-35 | 9
  Post booster 4, Day 21-35: number analyzed (Participants) | 10
  Post booster 4, Day 21-35 | 7
  Post booster 5, Day 21-35: number analyzed (Participants) | 3
  Post booster 5, Day 21-35 | 3
  Annual (11-13 months): number analyzed (Participants) | 48
  Annual (11-13 months) | 37
  Closeout: number analyzed (Participants) | 87
  Closeout | 75

2. Primary Outcome: Response Rates of Post Dose 2: Day 21-35 PRNT80 Titers
Description: Subject response rates for PRNT80 titers for post dose 2, days 21-35. The per-protocol population was used for immunogenicity analyses. Only subjects who were vaccinated according to the schedule defined in the protocol were included in the per-protocol population. Only observations or specimens collected according to the protocol were included in the analyses using the per protocol population. If a subject received one or more treatments out of compliance with the protocol schedule, any observations or specimens collected after the out-of-compliance treatment were excluded from the analyses using the per-protocol population.
Time Frame: Post dose 2, days 21-35
Population: Only observations or specimens collected according to the protocol were included in the analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination
Number analyzed (Participants) | 138
Participants
  Responders: number analyzed (Participants) | 41
  Responders: Year: 2008 | 8
  Responders: Year: 2009 | 4
  Responders: Year: 2010 | 10
  Responders: Year: 2011 | 12
  Responders: Year: 2013 | 5
  Responders: Year: 2014 | 2
  Non-responders: number analyzed (Participants) | 26
  Non-responders: Year: 2008 | 14
  Non-responders: Year: 2009 | 6
  Non-responders: Year: 2010 | 3
  Non-responders: Year: 2011 | 0
  Non-responders: Year: 2013 | 3
  Non-responders: Year: 2014 | 0

3. Primary Outcome: Response Rates of Pre-Month 6 PRNT80 Titers
Description: Subject response rates for PRNT80 titers of pre-month 6. The per-protocol population was used for immunogenicity analyses. Only subjects who were vaccinated according to the schedule defined in the protocol were included in the per-protocol population. Only observations or specimens collected according to the protocol were included in the analyses using the per protocol population. If a subject received one or more treatments out of compliance with the protocol schedule, any observations or specimens collected after the out-of-compliance treatment were excluded from the analyses using the per-protocol population.
Time Frame: Pre-month 6
Population: Only observations or specimens collected according to the protocol were included in the analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination
Number analyzed (Participants) | 138
Participants
  Responders: number analyzed (Participants) | 28
  Responders: Year: 2008 | 7
  Responders: Year: 2009 | 3
  Responders: Year: 2010 | 8
  Responders: Year: 2011 | 6
  Responders: Year: 2013 | 3
  Responders: Year: 2014 | 1
  Non-responders: number analyzed (Participants) | 33
  Non-responders: Year: 2008 | 13
  Non-responders: Year: 2009 | 6
  Non-responders: Year: 2010 | 4
  Non-responders: Year: 2011 | 4
  Non-responders: Year: 2013 | 5
  Non-responders: Year: 2014 | 1

4. Primary Outcome: Response Rates of Post Month 6: Day 21-35 PRNT80 Titers
Description: Subject response rates for PRNT80 titers for post month 6, days 21-35. The per-protocol population was used for immunogenicity analyses. Only subjects who were vaccinated according to the schedule defined in the protocol were included in the per-protocol population. Only observations or specimens collected according to the protocol were included in the analyses using the per protocol population. If a subject received one or more treatments out of compliance with the protocol schedule, any observations or specimens collected after the out-of-compliance treatment were excluded from the analyses using the per-protocol population.
Time Frame: Post month 6, days 21-35
Population: Only observations or specimens collected according to the protocol were included in the analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination
Number analyzed (Participants) | 138
Participants
  Responders: number analyzed (Participants) | 49
  Responders: Year: 2008 | 2
  Responders: Year: 2009 | 16
  Responders: Year: 2010 | 9
  Responders: Year: 2011 | 11
  Responders: Year: 2012 | 2
  Responders: Year: 2013 | 1
  Responders: Year: 2014 | 6
  Responders: Year: 2015 | 2
  Non-responders: number analyzed (Participants) | 11
  Non-responders: Year: 2008 | 0
  Non-responders: Year: 2009 | 8
  Non-responders: Year: 2010 | 1
  Non-responders: Year: 2011 | 1
  Non-responders: Year: 2012 | 0
  Non-responders: Year: 2013 | 0
  Non-responders: Year: 2014 | 1
  Non-responders: Year: 2015 | 0

5. Primary Outcome: Response Rates of Post Booster 1: Day 21-35 PRNT80 Titers
Description: Subject response rates for PRNT80 titers for post booster 1, days 21-35. The per-protocol population was used for immunogenicity analyses. Only subjects who were vaccinated according to the schedule defined in the protocol were included in the per-protocol population. Only observations or specimens collected according to the protocol were included in the analyses using the per protocol population. If a subject received one or more treatments out of compliance with the protocol schedule, any observations or specimens collected after the out-of-compliance treatment were excluded from the analyses using the per-protocol population.
Time Frame: Post booster 1, days 21-35
Population: Only observations or specimens collected according to the protocol were included in the analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination
Number analyzed (Participants) | 138
Participants
  Responders: number analyzed (Participants) | 82
  Responders: Year: 2008 | 34
  Responders: Year: 2009 | 23
  Responders: Year: 2010 | 11
  Responders: Year: 2011 | 3
  Responders: Year: 2013 | 6
  Responders: Year: 2014 | 3
  Responders: Year: 2015 | 2
  Non-responders: number analyzed (Participants) | 25
  Non-responders: Year: 2008 | 10
  Non-responders: Year: 2009 | 13
  Non-responders: Year: 2010 | 1
  Non-responders: Year: 2011 | 0
  Non-responders: Year: 2013 | 0
  Non-responders: Year: 2014 | 1
  Non-responders: Year: 2015 | 0

6. Primary Outcome: Response Rates of Annual (11-13 Months) PRNT80 Titers
Description: Subject annual response rates for PRNT80 titers for months 11-13. The per-protocol population was used for immunogenicity analyses. Only subjects who were vaccinated according to the schedule defined in the protocol were included in the per-protocol population. Only observations or specimens collected according to the protocol were included in the analyses using the per protocol population. If a subject received one or more treatments out of compliance with the protocol schedule, any observations or specimens collected after the out-of-compliance treatment were excluded from the analyses using the per-protocol population.
Time Frame: Months 11-13
Population: Only observations or specimens collected according to the protocol were included in the analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination
Number analyzed (Participants) | 138
Participants
  Responders: number analyzed (Participants) | 39
  Responders: Year: 2008 | 11
  Responders: Year: 2009 | 3
  Responders: Year: 2010 | 12
  Responders: Year: 2011 | 6
  Responders: Year: 2013 | 5
  Responders: Year: 2014 | 2
  Non-responders: number analyzed (Participants) | 14
  Non-responders: Year: 2008 | 4
  Non-responders: Year: 2009 | 6
  Non-responders: Year: 2010 | 0
  Non-responders: Year: 2011 | 2
  Non-responders: Year: 2013 | 2
  Non-responders: Year: 2014 | 0

7. Secondary Outcome: Number of Subject Experiencing Local and Systemic Adverse Events
Description: Number of subjects of who experienced and didn't experience local and systemic adverse events after vaccination and booster.
Time Frame: vaccination/booster days 0-28 for up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Vaccination - Primary; Vaccination - Booster: Inactivated, Dried, TSI-GSD 104, EEE
Arm/Group | Vaccination - Primary | Vaccination - Booster
Number analyzed (Participants) | 67 | 132
Participants
  No AEs: Male subjects | 19 | 47
  No AEs: Female subjects | 10 | 29
  Had AEs: Male subjects | 18 | 30
  Had AEs: Female subjects | 20 | 26

ADVERSE EVENTS:
Time Frame: vaccination and booster days 0-28 for up to 5 years
Groups:
- Vaccination/Booster: Inactivated, Dried, TSI-GSD 104, EEE
  Inactivated, Dried, TSI-GSD 104, EEE: Subjects will receive 0.5ml SQ, as a two-dose primary series (days 0 and 28) and 0.1ml, as a mandatory booster dose at 6 months. A booster dose may be administered before 6 months if PRNT80 is < 1:40 after day 28. Up to four booster doses may be given in any 1-year period.
Arm/Group | Vaccination/Booster
All-Cause Mortality (participants affected / at risk) | 0/136
Serious Adverse Events (participants affected / at risk) | 5/136
Other Adverse Events (participants affected / at risk) | 73/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccination/Booster (N=136)
Atrial febrillation (Cardiac disorders) | 1 (2)
Biscuspid aortic valve (Congenital, familial and genetic disorders) | 1 (1)
Viral pericarditis (Infections and infestations) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccination/Booster (N=136)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal destension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Allergic rhinitis (Immune system disorders) | 1 (1)
Amoebic dysentery (Gastrointestinal disorders) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bicuspic aortic valve (Cardiac disorders) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Chills (Musculoskeletal and connective tissue disorders) | 3 (3)
Colon cancer (Musculoskeletal and connective tissue disorders) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Diarrhea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 19 (19)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 21 (21)
Hyperhidrosis (General disorders) | 1 (1)
Injection site anaesthesia (General disorders) | 1 (1)
Injection site erythema (Injury, poisoning and procedural complications) | 16 (16)
Injection site haematoma (Injury, poisoning and procedural complications) | 10 (10)
Injection site induration (Injury, poisoning and procedural complications) | 5 (5)
Injection site pain (Injury, poisoning and procedural complications) | 12 (12)
Injection site paraesthesia (Injury, poisoning and procedural complications) | 1 (1)
Injection site pruritus (Injury, poisoning and procedural complications) | 9 (9)
Injection site swelling (Injury, poisoning and procedural complications) | 1 (1)
Injection site warmth (Injury, poisoning and procedural complications) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Middle ear infection (Ear and labyrinth disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 7 (7)
Oedema peripheral (Metabolism and nutrition disorders) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Oropharyngeal pain (Gastrointestinal disorders) | 15 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Sinus headache (Nervous system disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 15 (15)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vessel puncture site haematoma (Vascular disorders) | 1 (1)
Viral pericarditis (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No